CLINICAL TRIAL: NCT02874040
Title: Phase II Evaluating Endoresection of the Tumor Scar or Transpupillary Thermotherapy When Endoresection is Not Feasible After Proton Beam Therapy for the Treatment of Large Uveal Melanomas
Brief Title: Endoresection of the Tumor Scar or Transpupillary Thermotherapy for the Treatment of Large Uveal Melanomas (Endoresection-Laser)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC 2012-03
Record Dates: First submitted 2016-08-11; First posted 2016-08-22 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Uveal Melanoma; Melanoma, Uveal
MeSH Terms: conditions — Uveal Melanoma | interventions — Lasers, Semiconductor; Hyperthermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): endoresection of the tumor scar or, when surgery is not possible, transpupillary thermotherapy on the tumor scar
  Interventions: Procedure: Endoresection; Procedure: Laser diode

INTERVENTIONS:
Procedure: Endoresection — Endoresection of the tumor scar
Procedure: Laser diode — Transpupillary thermotherapy by laser diode on the tumor scar
  Other Names: Thermotherapy

SUMMARY:
Study the efficacy of endoresection of the tumor scar or, when surgery is not possible, transpupillary thermotherapy on the tumor scar to prevent neovascular glaucoma and secondary enucleation

ELIGIBILITY:
Inclusion Criteria:

* Tumor of 7 mm of thickness or more
* Patients treated by proton beam therapy
* Patients aged at least 18 years
* Patients clearly informed of the study, having received the letter of information and signed the consent

Exclusion Criteria:

* Massive extrascleral extension posterior to the equator
* Patients with metastasis at diagnosis.
* Patients with glaucoma before the radiation therapy
* Patients with opaque media preventing transpupillary thermotherapy
* Patients for whom follow up will be difficult due to geographical, social or psychological reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-04-19 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Post-treatment complication incidence. | 3 years
  observed complications are : Number of glaucomas, numbrer of retinal detachment and number of secondary enucleations.

SECONDARY OUTCOMES:
Measure of tumor scar thickness | 3 years
Toxicity and side effects evaluation according to NCI-CTCAE v4.0 scale | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie CASSOUX, MD, PhD, Study Director — Institut Curie
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: No